CLINICAL TRIAL: NCT05401006
Title: Evaluation of the Effect of Acitretin Versus Narrowband Ultraviolet B on Serum Neopterin Level in Psoriatic Patients .
Brief Title: Effect of Acitretin Versus Narrowband Ultraviolet B on Neopterin Level in Psoriatic Patients .
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Fatma Elsayed abd Elfatah Elsayed, Resident doctor, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 209/6/21
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Acitretin; Capsules

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acitretin (Active Comparator): Patients will Receive Acitretin (0.25-1 mg /kg/day )for 3months .
  Interventions: Drug: Acitretin 25Mg Cap
- Narrowband ultraviolet B (Active Comparator): Patients will receive Narrowband UVB( 3session /week ) for 3months.
  Interventions: Radiation: Narrowband ultraviolet B
- Combination of Narrowband ultraviolet B and Acitretin (Active Comparator): Patients will receive Acitretin (0.25-1 mg /kg/day ) and Narrowband UVB( 3session /week ) for 3 months.
  Interventions: Drug: Acitretin 25Mg Cap; Radiation: Narrowband ultraviolet B

INTERVENTIONS:
Drug: Acitretin 25Mg Cap — Acitretin is an oral retinoid (a derivative of vitamin A) given in a dose 0.25-1 mg /kg/day for 3months in psoriatic patients
  Arms: Acitretin; Combination of Narrowband ultraviolet B and Acitretin
Radiation: Narrowband ultraviolet B — Narrowband UVB is the most common form of phototherapy used to treat psoriasis, given 2-3 sessions per week for 3 successive months
  Other Names: Narrowband UVB
  Arms: Combination of Narrowband ultraviolet B and Acitretin; Narrowband ultraviolet B

SUMMARY:
To evaluate effect of acitretin versus Narrowband UVB on serum level of neopterin in psoriatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with psoriasis diagnosed clinically Aged (15-60).

Exclusion Criteria:

* Patient with history of skin cancer.
* Patient with history of photosensitivity.
* Pregnancy and lactation.
* Liver failure.
* Renal failure.
* Patient with psoriatic artheritis.
* Patient with allergy to product or any of its components.
* Patient with poorly controlled dyslipidemia.
* Patient receiving tetracyclines.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-05 (Actual); Primary Completion 2022-06-05 (Estimated); Study Completion 2023-06-05 (Estimated)

PRIMARY OUTCOMES:
Serum Neopterin in psoriasis | 3 Months
  Measurement of Neopterin in psoriatic patients before and after treatment with NB-UVB, Acitretin and combination of both modalities using ELISA (enzyme-linked immunosorbent assay).

SECONDARY OUTCOMES:
Treatment of psoriasis | 3 Months
  Clinical evaluation: Assessment of disease severity will be performed by using psoriasis area severity index (PASI score) before and after treatment with NB-UVB, Acitretin and combination of both modalities.

CONTACTS AND LOCATIONS:
Locations (1):
- South Valley University, Qina, Egypt